CLINICAL TRIAL: NCT03612440
Title: Effects of Dexmedetomidine on Oxygenation Index, Respiratory Index and Inflammatory Factors in Patients Undergoing Palatopalatyngoplasty
Brief Title: Effects of Dexmedetomidine on OI, RI and Inflammatory Factors in Patients Undergoing Palatopalatyngoplasty.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MHX07
Record Dates: First submitted 2018-06-19; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Adverse Effect
Keywords: dexmedetomidine; oxygenation index; respiratory index; inflammatory factors
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D (Experimental): 40 patients receive a loading infusion of dexmedetomidine (1ug/kg)for 20min follow by a maintenance infusion (0.4ug/kg/h) continued until the end of the surgery
  Interventions: Drug: dexmedetomidine
- Group C (Placebo Comparator): 40 patients receive matching placebo (normal saline)
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: dexmedetomidine — receive a loading infusion of dexmedetomidine (1ug/kg)for 20min follow by a maintenance infusion (0.4ug/kg/h) continued until the end of the surgery
  Arms: Group D
Other: normal saline — receive matching placebo (equal volum of normal saline)
  Arms: Group C

SUMMARY:
The purpose of this study is to investigate the efficacy of dexmedetomidine on oxygenation index, respiratory index and inflammatory factors, and to explore the protective effect of the dexmedetomidine on respiratory function in patients undergoing palatopalatyngoplasty.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome is common among people, especially among obese people, Which is characterized by periodic or complete upper airway obstruction and hypoxia during sleep. Intermittent hypoxia contributes to the lung damage by increased oxidative stress, inflammation. Some researchers suggested that dexmedetomidine can inhibit inflammatory reaction and lessen the damage of respiratory function. The aim of this study is to investigate the efficacy of dexmedetomidine on oxygenation index, respiratory index and inflammatory factors, and to explore the protective effect of the dexmedetomidine on respiratory function in patients undergoing palatopalatyngoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing palatopalatyngoplasty
* ASA physical status II-III
* Aged 18-65 years
* BMI 18.5-30kg/m2

Exclusion Criteria:

* Bradycardia
* Atrioventricular block
* Allergic to the drugs
* Complicating pulmonary disease(including pulmonary infection,COPD, asthma and so on)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
The Oxygenation Index | Intraoperative and immediately after surgery
  Arterial blood samples were sampled before anaesthesia induction and immediately after surgery for the oxygenation index by using blood gas analyzer.
The Respiratory Index | Intraoperative and immediately after surgery
  Arterial blood samples were sampled before anaesthesia induction and immediately after surgery for the respiratory index by using blood gas analyzer.

SECONDARY OUTCOMES:
Change of tumor necrosis factor-α before anesthesia and immediately after surgery | Intraoperative and immediately after surgery
  Blood samples were sampled before anaesthesia induction and immediately after surgery for the serum tumor necrosis factor-α，which were analyzed by using enzyme linked immunosorbent assay (ELISA).
Change of interleukin-6 before anesthesia and immediately after surgery | Intraoperative and immediately after surgery
  Blood samples were sampled before anaesthesia induction and immediately after surgery for the serum interleukin-6, which were analyzed by using enzyme linked immunosorbent assay (ELISA).
Change of interleukin-10 before anesthesia and immediately after surgery | Intraoperative and immediately after surgery
  Blood samples were sampled before anaesthesia induction and immediately after surgery for the serum interleukin-10, which were analyzed by using enzyme linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Li Na, Principal Investigator — General Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No
safety

REFERENCES:
- [Derived] Li N, Zhang Y, Yang F, Zhang H, Yu X, Lu K, Wang J, Ma H, Ni X. Effects of dexmedetomidine on oxygenation and inflammatory factors in patients undergoing uvulopalatopharyngoplasty: a prospective, randomized, placebo-controlled trial. Sleep Breath. 2023 Jun;27(3):1099-1106. doi: 10.1007/s11325-022-02711-1. Epub 2022 Sep 27. PMID 36166132